CLINICAL TRIAL: NCT01549808
Title: Early Mobilisation in Intensive Therapy
Brief Title: Early Mobilization in Intensive Therapy
Acronym: MIT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Zealand (Other)
Collaborators: Capital Region (Unknown)
Responsible Party: Principal Investigator, Anne Skafte, Nurse, Region Zealand
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIT ITA SLS 4141RH
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Critical Illness
Keywords: ADL; activities of daily living; level of function
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- group 2 (Experimental): Participants:
  100 patients will be included in the observation phase of this project, and another 100 in the intervention phase, according to the following criteria: Patients hospitalized in Unit 4141, at Rigshospitalet or ICU at Slagelse, who have been intubated for more than 48 hours, age ≥18, and after positive confirmation from relatives that the patient before the hospitalization was able to read and understand instructions.
  The research is divided in 3 phases:
  1. An 8 month observation phase.Current practice relatede to mobilize is measured.
  2. An 2 month implementation phase and third: an 8 month intervention phase. The effect is measured as the difference in the functional level between the observation phase and the intervention phase related to primary and secondary outcome.
  The effect of the intervention is described by using following test:
  walking distance,ADL function, capability to sit and stand
  Interventions: Other: mobilization

INTERVENTIONS:
Other: mobilization — The patients are mobilized according to the mobilization protocol. The training concist of balance, muscle strength and staying power. Before the mobilization the patients ability to mobilization is evaluated according to contradictions and pre screening (exh 2,3). The primary nurse and the physiotherapist evaluate and allocate patients to mobilization stage. All patients is mobilized minimum 3 times at day (exh 2) and is supported as a minimum of two persons. Before each activity the patient must have a rest period of ½ hour. The patients security during mobilization is registried (exh 1,3). The mobilization stops if patients security is affected. During walk patients is followed by a chair, in order to prevent or cushion a fall.
Other: mobilization — sitting, standing and walking

SUMMARY:
Abstract Many patients experience serious reduced functional ability after a critical illness and hospitalization in an Intensive Care Unit. The cause of the reduced functional ability is the combination of critical illness and immobilization following treatment with a ventilator. The functional ability of patients can be affected up till a year after the discharge, and may shows a decrease in ability to walk and in problems with focusing.

Studies show that it is safe and possible to mobilize the patients with for instance bed bikes, sitting up and standing up, even during ventilator therapy. The effect is shown as lesser days with delirium, on a ventilator therapy or hospitalization. No study has shown how early and at which intensity a patient can be mobilized. Our hypothesis is that an early systematic mobilization improves functional ability of the critically ill patient, mentally, physically and their life expectancy. The purpose of this study is to evaluate a mobilization protocol applied at critically ill patients, including a contribute related to knowledge of how soon and how intense patients ventilated for more than 48 hours can endure mobilization. To evaluate the connections between functional ability and life expectancy for critically ill patients are compared to a population matching in age.

This intervention project has a multicenter design with pre- and post research related to effect in early systematic mobilization of critically ill patients. 200 patients are included in the project.

Data are collected at tests showing the functional ability of patients in different ways. The tests are made at the discharge from the Intensive Care Unit and 5 days after at their wards and again at 3 and 12 month from discharge when the patients have returned to their home. The project started in February 2011 and is expected to end in May 2013, findings is expected in November 2013.

DETAILED DESCRIPTION:
Background Many patients experience serious reduced functional ability in form of physical and mental problems (1) after a critical illness and prolonged stay at an Intensive Care Unit. The critical illness entails the need for sedation and mechanical ventilation leading to immobilization as a consequence.

The combination of critical illness and immobilization leads to an increased risk of further muscle deterioration and it is assumed that this condition deteriorates the inflammatory response (2, 3, 4, 5).

Immobilization is an important contributory cause of reduced functional ability independent of critical illness. The deterioration is noticed up till a year after the discharge from hospital (1, 6) and physically it is shown in a reduced ability to walk (1, 6, 7), and mentally as delirium, associated with increased mortality and an extended period of hospitalisation. The mentally effects show a deterioration 1 year after the discharge from hospital.

The symptoms appear as difficulty concentrating and evaluated poor health (1, 6, 7).

Mobilization has a positive effect on the functional ability of patients, physically and mentally (8, 9, 10, 11, 12) even during mobilizing in connection with wake up calls of sedated patients 10). The patients experience less fear and dependency, they are in control to a greater extent (10) and also a significant increase in the ability to walk is shown (13). The mobilized patients have fewer days of delirium, mechanical ventilation and lesser days at Intensive Care Units (10, 12). It is possible to mobilize critically ill patients in bed by means of passive and active exercises. The exercises consist of getting out of bed, sitting on the edge of the bed, moving from bed to chair, standing on the floor, standing up, sitting in a chair and walking (10,13,14,15,16), but it is recommended that there is a close interdisciplinary collaboration between nurse and physiotherapist (17, 18, 19, 20, 21, 22).

Several studies (23, 24, 25, 26, 27, 28) show that it is safe and possible to mobilize critically ill patients while they receive mechanical ventilation. The incidence is less than 1 % (22) and is not directly related to age, sex, number of organ failure, co-morbidity or endo-tracheal tube (10, 21,22,25). The incidences appear as deceased SAT < 80 % (10, 17, 22, 24), subsidence of prostration without sustaining any damage (22), discontinuation of enteral feeding probe (22) or arterial catheter (10), changes in the systolic pressure (10,21,22), or patient-ventilator-asynchrony (10). It is recommended that the mobilization is structured (10, 15, 18, 22) by guidelines or protocols, and that the patients are screened before the mobilization. It is however not obvious, how soon and how intense patients can endure mobilizing.

Our hypothesis is that an early systematic mobilization improves the functional ability of critically ill patients, mentally and physically.

The purpose of this study is:

* To document the effects of early systematic mobilization of critically ill patients -
* to evaluate a mobilization protocol applied to critically ill patients, including a contribute related to knowledge of how soon and how intense patients can endure mobilization.
* To evaluate connections between functional ability and life expectancy of critically ill patients compared to a population matching in age.

The primary outcome is to measure the functional ability of the patients related to systematic mobilization. The patients stamina, balance, strength, experience and sense of control and emotional energy in relation to social contact is also measured. Correlation between functional ability and life expectancy is measured through their own judgment in relation to their physical level of activity, before hospitalisation and after discharge.

The secondary outcome is to measure mortality, days with mechanical ventilation, number of days of delirium, and bed rest at the Intensive Care Units and in the hospital, and factors contributing to critical illness which could influence the patients ability to recover (viewed as mobilization) are also measured.

Design and method:

This intervention project has a multicenter design with pre- and post research related to the effect of early systematic mobilization of critically ill patients (29).

Intervention and data collection:

The research is divided in 3 phases: An 8 month observation phase, a 2 month implementation phase and an 8 month intervention phase. The effect is measured as the difference in the functional level between the observation phase and the intervention phase related to primary and secondary outcome.

Phase 1: Observation phase The patients are mobilized according to the present routine of the hospital units without any guidelines. Data is registered on "the observation form" (exh1), and collected in the light of the present routine of the units. Before the form is used, the staff is instructed verbally and in writing.

Inter-observer variation is measured and tested at 8 nurses and by Kappa statistic. Acceptable values of Kappa are 0.61-0.80 corresponding to a high level of agreement.

Phase 2 implementation phase The mobilization protocol (exh 2) is formulated, inspired by Perme (15) and Gosselink (28) and in collaboration with physiotherapists at Slagelse Hospital, as a support for the staff during early systematic training. In order to strengthen the project, the staff is involved in the process early, when the mobilization protocol is used (31, 32). In both units there are established "steering groups" before the protocol is made. The staff is introduced to the protocol in this phase, and it is expected that the implementation is finished within a period of two month.

Phase 3 intervention phase The patients are mobilized according to the mobilization protocol. The training consists of improving the balance, muscle strength and stamina. Before the mobilization the abilities of the patients are evaluated according to contradictions and prescreening (exh 2, 3). The primary nurse and the physiotherapist evaluate and allocate patients to the best possible mobilization stage. All patients are mobilized minimum 3 times a day (exh 2) and the have the support of two persons as a minimum. Before each activity the patient must have a rest period of ½ hour. The security of the patients during mobilization is registered (exh 1, 3). The mobilization stops if the security is affected. During walks patients are followed by a member of staff pushing a chair behind them, in order to prevent or cushion a fall.

Participants:

100 patients will be included in the observation phase of this project, and another 100 in the intervention phase, according to the following criteria: Patients hospitalized in Unit 4141, at Rigshospitalet or ICU at Slagelse, who have been intubated for more than 48 hours, age ≥18, and after positive confirmation from relatives that the patient before the hospitalization was able to read and understand instructions.

Excluded:

Patients with a terminal illness, users of wheelchairs, patients with a known cognitive disturbance, open thorax, ECMO, VAD, IABP, and patients where mobilization is contradicted, and finally patients living outside Sjaelland, Lolland and Falster.

Patients vary from being totally dependent of help towards an alteration of independence and this requires a method to measure which can detect the shift in their functional ability during hospitalization and after discharge from the hospital. No single method of measurement detects this shift per se and it is therefore necessary to use various methods to measure the functional ability of the patients.

The appraisal of the mental ability of patients, understood as consciousness is evaluated daily with RASS score, and delirium through CAM ICU (exh 1, 3).

After discharge the patients evaluate their own functional ability, understood as control and emotional energy related to social contact with other human beings, in the questionnaire SF 36 (exh 4). All 3 measurements are validated in a number of International and Danish projects and are therefore regarded as suitable for critically ill patients (34, 35) The appraisal of the functional ability of patients, understood as the capability to mobilize during hospitalization is "the Cumulated Ambulation Score" (CAS). CAS shows the independency and development of the patients regarding the basic mobility in days, understood as capability to get out of bed, to stand, to sit and to walk (exh 1, 3). CAS, which originally was validated for patients with hip fractures, has been recommended for a broader group of patients (36). Pain is evaluated through a numeric rang scale (NRS) (37) before mobilization (exh 1, 3). In addition the varying forms of mobilization like standing up, sitting down, walking and also accidents are registered (exh 1,3) At discharge from the ICU to a ward or their own home, the development in functional ability is registered by means of ADL, Bartel-20 (exh 5). ADL registration shows the ability of patients to fulfill daily living, Bartel-20 clarifies the functional ability in 10 selected areas (38, 39) and is validated both internationally and in Denmark (40). In order to follow the development of the physical strength, endurance and balance the "Rejse Sætte Sig" test is used (exh 6) and also "Timed Up and Go" (TUG) (exh 7). The test "Rejse Sætte Sig " clarifies the level of strength in the lower part of their bodies, their balance and risk of falling. The TUG test is recommended to predict the physical strength and balance of patients who are neither self-reliant nor totally dependent (41).

The shift in the ability of patients to be self-reliant at home is evaluated in "New Mobility Score" (exh 8). The test which clarifies the ability to be self-reliant at home shows an acceptable reliability score (42, 43, 44).

In order to measure connections between the functional ability and life expectancy matched to the Danish population and correlating in age "Fysisk Aktivitet i Fritiden" is used (exh 9). The score which clarifies the physical activities is also recommended to clarify the risk of dependency and death (45).

In order to estimate the outcome of critically ill patients Apache and SAPS are used. Both are validated for critically ill patients (46, 47).

Statistic Calculation of strength is done based on previous studies and the key parameters are walking distance in meter and ADL measured in bartel-20.

Sample size calculation for ADL Interval scale Type 1 errors: 5% Est.SD:43 The least difference between mean: 20,00 Type 2 errors: 20% Patients needed both group: 72 Sample size calculation for walking distance (20 m estimate) Interval scale Type 1 errors: 5% Est.SD: 20 The least difference between mean: 10, 00 Type 2 errors: 20% Patients needed both group: 62

Processing of data:

Data are registered in Excel, processed in SPSS and statistically compared X2 ((48) and kept safe in servers with "log on" and back ups, at Rigshospital and Slagelse Hospital, and are only accessible for members of the project group.

Timeschedule The research started at 2011.02.01. The observation phase runs from 2011.02.01 to 2011.12.31. The implementation phase starts 2012.01.01 and is expected to end the 2012.03.31. The intervention phase is scheduled when the mobilization protocol is implemented, probably in 2012.04.01. The last patient is expected to be included in Jan 2013. The research is expected to end 2014.01.31 Preliminary results are expected in Apr. 2014. Final results are expected in July 2014.

Settings The Anesthesiological Thorax ICU (4141) at Rigshospitalet has room for 19 patients. The most commonly treated problems are heart failure, thorax surgery, lung transplantation and thoracotomy. Adverse side effects are circulation failure, renal failure or sepsis with a need for gradual reduction from ventilator and physical rehabilitation. The ICU has single rooms, double rooms, one room for four patients and one for six patients. The physiotherapist evaluates and starts the training which consists of excises to improve strength, the ability to sit down, to stand up and to walk. The training is always medically prescribed. The different transitions are taking place by use of a lift.

ICU at Slagelse Hospital has room for 10 patients, all in single rooms. The most commonly treated patient groups are patients with complications after gastointestinal surgery, medical or orthopedic patients. Compared to 4141 at Rigshospitalet the ICU at Slagelse also treats patients with adverse side effects as circulation failure, renal failure, sepsis or patients with a need for gradual reduction from a ventilator and need of physical rehabilitation. As in 4141 at Rigshospitalet the physiotherapy is medically prescribed. The training consists of prevention when the patient can not move, and when the patient can cooperate the training consists of improving the physical functions, such as moving around in the bed, sitting at the bedside, standing up, turning around and walking. As in 4141 at Rigshospitalet the different transitions are taking place by use of a lift in the ceiling at the beginning. The assistive technology used in both units, are ceiling lifts, walkers, wheelchairs, adaptable armchairs and mobile ventilators.

Processing of data:

In the observation phase and in the intervention phase data are collected as follows: The nurse who is caring for the patient every day collects data regarding the evaluation of consciousness, pain, basic mobility and security during mobilization.

A member of the project group (exh 12) includes the patient and obtains consent, and is performing the test at discharge from the ICU, and again on the 5th day at the ward, and finally at home after discharge. Before the visit at home, the patient is contacted by telephone in order to accept and schedule a date for the visit and to allow us to send out a questionnaire. The tests are conducted as close as possible to the day for discharge from the ICU, the 5th day at the ward and 3 and 12 month after returning home. Deviation from the exact date can for the first 2 tests vary +/- 1 day, and for the test after 3 and 12 month +/- 10 days.

Ethics The project is approved by "The Science/Ethical Committee" (exh 13) and the "Datatilsynet" according to the "Law of Privacy", and the data are stored according to regulations from the "Datatilsynet" (exh 14). The project is carried out according to "Ethical Guidelines for Research performed by Nurses in the Nordic Area", building on "Ethical Principles" expressed in the Helsinki Declaration and UN Human Rights Declaration (49, 50).

In the observation phase, approval is gathered as soon as the patient is regarded as being clear minded. If the patient is not situated in a single room, and because it is not always possible or save to move the patient out of the bedroom, approval, in both the observation phase and in the intervention phase, will be obtained with regard to the integrity of the patient. The participants will be informed equally verbally and in writing and with the present of a relative. If a participant does not wish to continue the project, he will be excluded promptly.

In the intervention phase the participants are often sedated and therefore it is necessary to inform a relative/substitute/personal doctor both verbally and in writing in order to obtain the approval. The relative will be contacted by one of the members of the project group when the patient has been at the ICU for 24 hours, and approval is needed after further 24 hours. The verbal information will be giving by a member of the steering group in a separate room away from other patients. The written information will be handed out at the same time. Final approval will be requested, only when the written information has been read. As soon as the participant is assessed to be awake and clear minded, he will be asked for further participation.

Financing The results will be financed through the ICU accounts, but also by application to funds (exh 8,19).

Publication Results from the research, positive as well as negative, will be published in scientific journals and an application for an article in CCN will be made.

ELIGIBILITY:
Patients who will be included:

* Patients hospitalized in Unit 4141, at Rigshospitalet or ICU at Slagelse, who have been intubated for more than 48 hours,
* age ≥ 18, and
* after positive confirmation from relatives that the patient before the hospitalization was able to read and understand instructions.

Patients who will be excluded:

* Patients with a terminal illness,
* users of wheelchairs,
* patients with a known cognitive disturbance,
* open thorax,
* ECMO,
* VAD,
* IABP,
* patient who is not allowed to mobilizing during their stay in ICU, and finally
* patients living outside Sjaelland, Lolland and Falster.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-01 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to measure the functional ability of the patients | 3 years
  The primary outcome is to measure the functional ability of the patients related to systematic mobilization. The patients stamina, balance, strength, experience and sense of control and emotional energy in relation to social contact is also measured. Correlation between functional ability and life expectancy is measured through their own judgment in relation to their physical level of activity, before hospitalisation and after discharge.

SECONDARY OUTCOMES:
Is to measure the effect of mobilization related to time in hospital | 2. year
  The secondary outcome is to measure mortality, days with mechanical ventilation, number of days of delirium, and bed rest at the Intensive Care Units and in the hospital, and factors contributing to critical illness which could influence the patients ability to recover (viewed as mobilization) are also measured.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Skafte, Nurse, Principal Investigator — Slagelse Sygehus, Danmark
Locations (1):
- Slagelse Sygehus, intensiv afdeling, Slagelse, Denmark